CLINICAL TRIAL: NCT04526145
Title: Operating Under Resilience (OUR) Project: Stress and Emotion Management for Black/African American Women With Hypertension In a Covid--19 Social Distancing Society
Brief Title: OUR Stress/ Emotion Management for Black/African American Women With Hypertension
Acronym: OUR-Project
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University (Other)
Responsible Party: Principal Investigator, Kathy D. Wright, Assistant Professor, Ohio State University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 2020B0182
Record Dates: First submitted 2020-08-10; First posted 2020-08-25 (Actual); Results first posted 2025-05-16 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Stress, Psychological
Keywords: hypertension; Covid-19; Black and African American women; Mindfulness; Diet
MeSH Terms: conditions — Stress, Psychological; Hypertension; COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Stress and emotion Management for Black/African Americ (Experimental): Four weekly sessions delivered in a group format via Zoom teleconference. The following topics are listed in the workbook: Planning Your Information Diet; My Spheres of Influence Worksheet; Practical Wisdom for Tolerating Uncertainty; Reducing Anxiety With Thought Challenging; Reducing Anxiety Through Distraction Activities; Starting a Planning Practice; Starting a Daily Gratitude Practice; Starting a Daily Breathing Practice; Improving the Quality of Your Social Connections; Developing a Regular Exercise Routine; and Creating Your Stress-Resilience Action Plan. Each session will begin with a 15-30 minute check in on what went well, challenges, and Coronavirus Anxiety workbook. The Coronavirus Anxiety Workbook topics are complementary and the sessions will tie together the themes of comprehensive stress and emotional management through blood pressure knowledge/self-monitoring, diet, interpersonal communication skills building, and sleep hygiene.
  Interventions: Behavioral: Stress and emotion management

INTERVENTIONS:
Behavioral: Stress and emotion management — Group intervention led by a nurse and dietitian to address stress, emotion management and healthy lifestyle for African American women with hypertension. The weekly sessions will include:how to manage stress during Covid-19, taking blood pressure, interpersonal relationships skills, mindful awareness, restful sleep, physical activity, and healthy eating.

SUMMARY:
Covid-19 is an additional stressor Black women have to deal with that may interfere with hypertension self-care management. Social connectedness is a source of resilience for Black women to promote mental and physical health. Unfortunately, in the face of the Covid-19 pandemic, social distancing is a challenge further isolating Black women from their networks. How is social connectedness to manage stress and emotional well-being in a social-distancing society for Black women with hypertension? The research team proposed a synchronous web-based version of Enhanced Co-Created Health Education InterventioN (eCo-CHIN) that build the success and best practices derived from the original intervention. A Covid-19 session will be included as a way of helping Black women to maintain resilience and self-care during stressful times. The eCo-CHIN intervention is innovative and timely because the research team are using a synchronous platform preparing Black women on how to deal with Covid-19 while taking care of self. The primary investigator for this pilot study (Dr. Wright) is a Black Early Stage Investigator and former KL2 (career development) awardee. The interdisciplinary research team has the expertise and resources to deliver this Enhanced Co-CHIN intervention.

DETAILED DESCRIPTION:
The rationale for the study is that the adherence to healthy self-care behaviors reduces poor nutrition, altered sleep, sedentary behavior, psychosocial stress, and emotional dysregulation, thereby reducing negative impacts on the brain, since all these factors contribute to neural inflammation and increased BP. Health-promoting self-care behaviors have the known short-term effect of enhanced cognitive function (processing speed, attention, and executive function) through the use of The Repeatable Neuropsychiatric Battery (RBANS) which is also an innovative component of OUR Project. Thirty middle-aged Black women (45-65 years old) with a self-reported diagnosis of hypertension will be enrolled. The development of this group-delivered intervention will be an iterative process, and the research team will use this pilot data to submit an R21 for a 12-week intervention through the National Institutes on Aging.

ELIGIBILITY:
Inclusion Criteria:

* English speaking,
* self-identification as Black/African America
* diagnosis of hypertension (treated with medications and or lifestyle management)
* female sex
* access to a smart phone or a computer capable of connecting to the Internet

Exclusion Criteria:

* no access to computer with internet Smart phone
* diagnosis of resistant hypertension defined as blood pressure that remains above goal despite concurrent use of three antihypertensive agents of different classes, one of which should be a diuretic/water pill.

Min Age: 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Self-report of female sex at birth.
Enrollment: 16 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2024-11-30 (Actual); Study Completion 2024-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kathy D Wright, PhD, RN, Principal Investigator — Assistant Professor
Locations (1):
- The Ohio State University, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 2 Consented individuals did not begin the study due to a change in eligibility prior to beginning of study.
Period: Overall Study
Arm/Group | Stress and Emotion Management for Black/African Americ
Started | 14
Completed | 9
Not Completed | 5
Not completed — Withdrawal by Subject | 5

BASELINE CHARACTERISTICS:
Arm/Group | Stress and Emotion Management for Black/African Americ
Number analyzed (Participants) | 14
Age, Customized [Count of Participants; unit: Participants]
  47-53 | 5
  54+ | 9
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 14
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 14
Years of Education [Count of Participants; unit: Participants]
  10+ | 14
  7-9 | 0
  0-6 | 0

OUTCOME MEASURES:

1. Primary Outcome: Determine the Feasibility of a Synchronous Web-based Health Education Program, of OUR Project.
Description: Weekly participant attendance will be recorded as date, month and year.
Time Frame: 4 weeks
Population: 4 weekly sessions, attendance at each session was measured
Measure: Mean (Standard Deviation); unit: weeks attendance/month
Arm/Group | Stress and Emotion Management for Black/African Americ
Number analyzed (Participants) | 14
weeks attendance/month | 2.93 (1.21)

2. Primary Outcome: Determine the Acceptability of a Synchronous Web-based Health Education Program, of OUR Project.
Description: Investigator generated questions regarding the acceptability of the program. There are 13 questions ranked on a 10 point scale, with higher scores indicating a stronger acceptability of the program. Total scores range from 13 to 130 for each individual. All scores are averaged.
Time Frame: 1 month and 6 months post intervention
Population: Some participants did not participate in the intervention acceptability testing.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Stress and Emotion Management for Black/African Americ
Number analyzed (Participants) | 7
score on a scale
  1 month post intervention | 98.6 (10.1)
  6 months post intervention | 96.1 (14.4)

3. Primary Outcome: Change From Baseline at 1 Month Weight.
Description: Weight measured in pounds.
Time Frame: Baseline to 1 month post baseline
Population: 5 participants were lost to follow up.
Measure: Mean (Standard Deviation); unit: pounds
Arm/Group | Stress and Emotion Management for Black/African Americ
Number analyzed (Participants) | 14
pounds
  Baseline | 234.3 (47.4)
  Post -1 Month: number analyzed (Participants) | 9
  Post -1 Month | 250.8 (50.9)

4. Primary Outcome: Change From Baseline at 1 Month Waist Circumference.
Description: Waist circumference measured in inches.
Time Frame: Baseline to 1 month post baseline
Population: 1 participant did not have waist circumference measured at baseline.
Measure: Mean (Standard Deviation); unit: inches
Arm/Group | Stress and Emotion Management for Black/African Americ
Number analyzed (Participants) | 13
inches
  Baseline | 44.5 (5.0)
  Post 1-Month: number analyzed (Participants) | 9
  Post 1-Month | 45.9 (6.9)

5. Primary Outcome: Change From Baseline at 1 Month Systolic Blood Pressure.
Description: Self-blood pressure collection using an automatic home blood pressure monitor systolic blood pressure in mmHg
Time Frame: Baseline to 1 month baseline
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Stress and Emotion Management for Black/African Americ
Number analyzed (Participants) | 13
mmHg
  Baseline | 128.5 (17.4)
  Post 1-Month | 122.5 (16.2)

6. Primary Outcome: Change From Baseline at 1 Month Diastolic Blood Pressure.
Description: Self-blood pressure collection using an automatic home blood pressure monitor diastolic blood pressure in mmHg
Time Frame: Baseline to 1 month baseline
Population: 1 participant did not have blood pressure measured at baseline
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Stress and Emotion Management for Black/African Americ
Number analyzed (Participants) | 13
mmHg
  Baseline | 87.0 (10.3)
  Post 1-Month | 83.4 (4.6)

ADVERSE EVENTS:
Time Frame: 3 month period post baseline
Description: Any untoward or unfavorable medical occurrence in a participant, including any abnormal sign (for example, abnormal physical exam or laboratory finding), symptom, or disease, temporally associated with the participant's participation in the research, whether or not considered related to the participant's participation in the research.
Arm/Group | Stress and Emotion Management for Black/African Americ
All-Cause Mortality (participants affected / at risk) | 0/16
Serious Adverse Events (participants affected / at risk) | 0/16
Other Adverse Events (participants affected / at risk) | 0/16

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-10-01): https://cdn.clinicaltrials.gov/large-docs/45/NCT04526145/Prot_SAP_000.pdf
  • Informed Consent Form (2021-10-01): https://cdn.clinicaltrials.gov/large-docs/45/NCT04526145/ICF_001.pdf